CLINICAL TRIAL: NCT04776200
Title: Mental Health Status of Women Who Attending Classical Ballet Dance
Brief Title: Classical Ballet Dance as a Recreational Activity for Adults Women
Status: Completed | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, ZEYNEP BAHADIR AGCE, Assistant Professor, Uskudar University
Other Study IDs: 61351342/2020-135
Record Dates: First submitted 2021-02-20; First posted 2021-03-01 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Occupational Therapy
Keywords: Dancing; occupational therapy; mental health; adults
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ballet Groups: It was invited the individuals, who were ongoing for at least 3 months in classical ballet dance activity in the dance studio, between December 2019 and March 2020.
- Control Groups: It was invited the individuals, who have just registered for classical ballet dance activity.

SUMMARY:
Classical ballet dance has just used therapeutically in recent years and can be a good recreational activity option at occupational therapy. The purpose of this study was to investigate whether participation in classical ballet dance activity for at least 3 months is associated with psychological distress, depression, anxiety, and well-being.

DETAILED DESCRIPTION:
A total of 128 adults participated in the study, sixty-four for Ballet Group (BG) and Control Group (CG). The psychological distress of the participants were evaluated with the Distress Tolerance Scale (DTS), anxiety and depression evaluated with Hospital Anxiety and Depression Scale (HADS), and well-being and quality of life evaluated with the World Health Organization Well-Being Index (WHO-5).

ELIGIBILITY:
Inclusion Criteria:

The ballet group's inclusion criteria

* age between 18 and 65 years,
* weekly attendance at ballet classes for at least 3 months

The control group's inclusion criteria

* age between 18 and 65 years,
* did not participate in any ballet activity.

Exclusion Criteria:(for both groups)

* Being a professional dancer or athlete
* Diagnosed with systemic diseases such as rheumatoid arthritis, diabetes
* Diagnosed with psychiatric disorders such as depression, anxiety

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Accepts Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
The World Health Organisation's Five Well-Being Index | 5 minutes. Each participant who meets the inclusion criteria was asked to fill out the form only once in beginning of the study.
  The World Health Organisation's Five Well-Being Index (WHO-5), which is developed by Bench et al., is a valid instrument for the psychometric evaluation of emotional well-being, and quality of life for the previous two weeks (Bech et al., 1996). This measure consists of 5-items, which respondents rated on a scale of "0- never" to "5- all the time". The WHO-5 low score "0" representing the worst possible well-being and "100" the best. The score of lower than 13 could be regarded as indicates poor quality of life.

SECONDARY OUTCOMES:
The Distress Tolerance Scale | 7 minutes.Each participant who meets the inclusion criteria was asked to fill out the form only once in beginning of the study.
  The Distress Tolerance Scale (DTS) is a 15- item, self-report used to assess psychological distress, which is developed by Simons and Gaher (Simons and Gaher, 2005).DTS was used as a function of the time period during which these data were collected. While the original scale has 4 factors Turkish version has 3 factors across Tolerance, Regulation, Self-Efficacy. 5-point Likert-type scale score changes between 1 strongly agree and 5 strongly disagree. The higher scores indicating higher psychological distress tolerance.
The Hospital Anxiety and Depression Scale | 10 minutes. Each participant who meets the inclusion criteria was asked to fill out the form only once in beginning of the study.
  The Hospital Anxiety and Depression Scale (HADS), which is developed by Zigmond et. all is a self-assessment tool for to use of detecting depression and anxiety (Zigmond and Snaith, 1983). HADS investigates how people have felt in the past week. It has included 14- items, which rated on a four-point scale and scored from 0-3, and two subscales, as anxiety (7 items) and depression (7 items), each part scores ranged from 0 to 21. Scores between 0 and 7 indicate normal emotional stated, and higher than 7 on the subscales of the HADS indicated anxiety and depressive disorder.

CONTACTS AND LOCATIONS:
Overall Officials: ZEYNEP BAHADIR AGCE, PHD, Study Director — occupational therapy
Locations (1):
- Zeynep Bahadır Ağce, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] da Costa ALB. (2012) Circle dance, occupational therapy and wellbeing: the need for research. British Journal of Occupational Therapy 75: 114-116.
- [Background] Houston S and McGill A. (2011) English National Ballet dance for Parkinson's: An investigative study. Report retrieved from: http://www. ballet. org. uk/media/filer_public/2015/08/20/english_ national _ballet_dance_ for_parkinsons_an_investigative_study. pdf on 6: 2016